CLINICAL TRIAL: NCT05140525
Title: Effects of Combination Medical Therapy Followed by Balloon Pulmonary Angioplasty on Right Ventricular-PA Coupling and Hemodynamics in Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Effects of Combination Medical Therapy Followed by BPA on Right Ventricular-PA Coupling and Hemodynamics in CTEPH
Acronym: EPIPHANY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Sudarshan Rajagopal (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor-Investigator, Dr Sudarshan Rajagopal, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105903
Record Dates: First submitted 2021-10-28; First posted 2021-12-01 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-06

CONDITIONS: CTEPH
Keywords: Inoperable; Post-PTE
MeSH Terms: interventions — macitentan; riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- participants with inoperable CTEPH (Active Comparator): subject with inoperable Chronic thromboembolic Pulmonary Hypertension
  Interventions: Drug: Macitentan Tablets; Drug: Riociguat; Device: balloon pulmonary angioplasty
- post PTE residual CTEPH (Active Comparator): Subject with post pulmonary endarterectomy (PTE) residual Chronic Thromboembolic Pulmonary Hypertension
  Interventions: Drug: Macitentan Tablets; Drug: Riociguat; Device: balloon pulmonary angioplasty

INTERVENTIONS:
Drug: Macitentan Tablets — 10 mg oral once daily
  Other Names: OPSUMIT
Drug: Riociguat — 1 mg to 2.5mg oral three times daily
  Other Names: Adempas
Device: balloon pulmonary angioplasty — on hemodynamics and RV function (including advanced assessments of RV-PA coupling

SUMMARY:
The main goal of this study is to determine the effects of combination medical therapy (Riociguat and Macitentan) and balloon pulmonary angioplasty (BPA) on hemodynamics and right ventricular (RV) function (including advanced assessments of RV-pulmonary artery (PA) coupling from invasive hemodynamics) in participants with inoperable or post-PTE residual CTEPH.

DETAILED DESCRIPTION:
Recent presented but unpublished results from trials of BPA vs riociguat for inoperable CTEPH (NCT02634203) have demonstrated that BPA provides a more significant hemodynamic benefit than medical therapy. The investigators hypothesize that participants who are treated with upfront combination medical therapy followed by BPA will have significant improvements in their hemodynamics and RV-PA coupling that can be monitored over time.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Age ≥ 18 years' old
2. Diagnosis of CTEPH
3. Not a candidate for PTE
4. Candidate for BPA based on suitable anatomy and disease burden
5. Treatment-naïve (no CTEPH or pulmonary arterial hypertension (PAH)-specific medical therapies) with plans for initiation of CTEPH/PAH-specific medical therapy and treatment with BPA.
6. Willing and able to give informed consent and adhere to visit/protocol schedules (Consent must be given before any study procedures are performed).

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the trials:

  1. Moderate to severe heart disease (LVEF < 45% or severe LV Hypertrophy)
  2. Sarcoidosis
  3. Active cancer
  4. Sickle cell anemia
  5. Liver disease (Childs-Pugh class C)
  6. Prisoners
  7. Pregnant, planning pregnancy or lactating
  8. Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine)
  9. Contraindication to riociguat or macitentan
  10. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in end-systolic elastance (Ees) divided by arterial elastance (Ea) (Ees/Ea) at three time points: Baseline, Timepoint 1 and Timepoint 2. | Baseline (before starting all treatments); Timepoint 1 (after starting medical therapy; up to 6 months after baseline); Timepoint 2 (after balloon pulmonary angioplasty (BPA); up to 12 months after baseline)
  Ees is a measure of right ventricular (RV) - pulmonary arterial (PA) coupling, with a normal value of Ees/Ea > 0.8 (dimensionless - no units). For subjects with Ees/Ea > 0.8 at the start of the study, we will evaluate the absolute change in Ees/Ea between timepoints. For those with an Ees/Ea < 0.8, we will also determine whether participants have an improvement to > 0.8.

SECONDARY OUTCOMES:
Change in six-minute walk distance (6MWD) in meters. | Baseline (before starting all treatments); Timepoint 1 (after starting medical therapy; up to 6 months after baseline); Timepoint 2 (after balloon pulmonary angioplasty (BPA); up to 12 months after baseline)
  6MWD will be determined at baseline, timepoint 1 and timepoint 2. Absolute change between these timepoints will be determined.
Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) in picogram/milliliters. | Baseline (before starting all treatments); Timepoint 1 (after starting medical therapy; up to 6 months after baseline); Timepoint 2 (after balloon pulmonary angioplasty (BPA); up to 12 months after baseline)
  NT-proBNP will be determined at baseline, timepoint 1 and timepoint 2. Absolute change between these timepoints will be determined.
Change in Cardiac index as measured by liters per minute per meters squared at right heart catheterization. | Baseline (before starting all treatments); Timepoint 1 (after starting medical therapy; up to 6 months after baseline); Timepoint 2 (after balloon pulmonary angioplasty (BPA); up to 12 months after baseline)
  Right heart catheterization will be performed at baseline, timepoint 1 and timepoint 2 and parameters determined. Absolute change between these timepoints will be determined.
Change in pulmonary vascular resistance as measured by Wood units at right heart catheterization. | Baseline (before starting all treatments); Timepoint 1 (after starting medical therapy; up to 6 months after baseline); Timepoint 2 (after balloon pulmonary angioplasty (BPA); up to 12 months after baseline)
  Right heart catheterization will be performed at baseline, timepoint 1 and timepoint 2 and parameters determined. Absolute change between these timepoints will be determined.
Change in right atrial pressure as measured by millimeters of mercury at right heart catheterization. | Baseline (before starting all treatments); Timepoint 1 (after starting medical therapy; up to 6 months after baseline); Timepoint 2 (after balloon pulmonary angioplasty (BPA); up to 12 months after baseline)
  Right heart catheterization will be performed at baseline, timepoint 1 and timepoint 2 and parameters determined. Absolute change between these timepoints will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Rajagopal, MD, PhD, Principal Investigator — Duke Health System
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No